CLINICAL TRIAL: NCT05477459
Title: Efficacy and Safety of Minidosing Lysergic Acid Diethylamide (LSD) for Chronic Cluster Headache: a Randomized Placebo-controlled Study
Brief Title: LSD to Improve Cluster Headache Impact Trial
Acronym: LICIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Canisius-Wilhelmina Hospital (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 131-2022
Record Dates: First submitted 2022-07-05; First posted 2022-07-28 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Chronic Cluster Headache
Keywords: Chronic cluster headache; Lysergic acid diethylamide
MeSH Terms: conditions — Cluster Headache | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: 3-week double-blind placebo-controlled intervention study, preceded by a 4-week baseline observation period and followed by 5 weeks post-treatment observation period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug or placebo are similar in appearance, taste and smell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Lysergic diethylamide tartrate (equivalent to 25 microgram LSD base), one dose every 3 days for 3 weeks (totalling 7 vials)
  Interventions: Drug: LSD tartrate
- Placebo (Placebo Comparator): Placebo vial looking like verum vial, one vial every 3 days for 3 weeks (totalling 7 vials)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LSD tartrate — LSD tartrate equivalent to 25 microgram LSD base
  Other Names: Lysergic acid diethylamide
  Arms: Verum
Drug: Placebo — Placebo with equal appearance
  Arms: Placebo

SUMMARY:
This study aims to investigate the efficacy and safety of LSD 25μg every 3 days for 3 weeks versus placebo in the treatment of chronic cluster headache (cCH).

It is a 3-week double-blind placebo-controlled intervention study, preceded by a 4-week baseline observation period and followed by a 5-week post-treatment observation period.

Primary objective: to evaluate the efficacy of LSD 25μg every 3 days for 3 weeks in cCH.

Additional objectives:

* To evaluate the safety of LSD 25μg every 3 days for 3 weeks in cCH.
* To explore the exposure-response relationship of 25μg LSD in cCH.
* To explore cost-effectiveness of treatment with LSD in cCH.
* To evaluate the efficacy of LSD on health-related quality of life.

DETAILED DESCRIPTION:
Treatment of cluster headache consists of acute remedies for attacks (mainly 100% O2, sumatriptan), transitional treatment for temporary frequency reduction (subcutaneous steroid injection at the greater occipital nerve (GON block), oral steroids or frovatriptan) and prolonged prophylaxis (e.g. verapamil, lithium, topiramate). Although the latter compounds have shown some efficacy in reducing the attack frequency, the evidence for their effect is weak. All current prophylactics are prescribed off-label and are limited in their utility due to associated side effects. Despite treatment, many (notably chronic) cluster headache patients continue suffering headache attacks.

Invasive, expensive treatments like hypothalamic deep brain stimulation, occipital nerve stimulation and sphenopalatine ganglion stimulation are last resort options. Recently, a monoclonal antibody targeting calcitonin gene related peptide (CGRP) received FDA approval for episodic cluster headache, but was shown to be ineffective in cCH. Thus, there is a considerable unmet need for effective treatments that are better tolerated, safe and affordable.

In this study, the investigators will assess the efficacy of prophylactic treatment with LSD in cCH. The evidence for the efficacy of LSD is limited, with the majority of data originating from case reports or uncontrolled and retrospective (internet) surveys. Nevertheless, these studies do provide indications that LSD may hold potential as a cluster headache prophylaxis.

The primary objective of this randomized double-blind placebo-controlled trial is to compare the efficacy of LSD 25μg every 3 days for 3 weeks versus placebo in cCH. The investigators aim to show that, at the end of treatment, verum is more efficacious than placebo with comparable tolerability in an ambulatory setting. To explore the sustainability of benefit the investigators will also assess the (sustained) response at 5 weeks post-treatment (8 weeks postrandomization).

If the study findings are positive, LSD should be further studied before use in routine clinical practice. Non-hallucinogenic low-dosed LSD may provide an alternative or adjunctive option for patients who do not respond to or cannot tolerate currently available treatments.

ELIGIBILITY:
Inclusion Criteria:

* CCH according to the International Classification of Headache Disorders version 3 (ICHD-3)
* At screening: stable weekly attack frequency in the 4 weeks prior to screening (assessed retrospectively), averaging at least 8 per week and each week within a 40% window around the average
* At randomization: average of at least 8 attacks per week and no absence of attacks on more than two consecutive days during baseline

Exclusion Criteria:

* Use of excluded concomitant treatment at screening (lithium; other prophylactics if not on a stable dose for less than one month; steroids/GON block within 2 months before screening; sphenopalatinum block, neurostimulation (changed setting within 3 months before screening) or botulinum toxin within 3 months before screening) and during the double-blind phase
* Use of LSD(-derivatives) (other than investigational drug), psilocybin, ketamine or cannabis within 3 months prior to screening and throughout the study
* Lifetime and/or family history (first degree relatives) of psychotic or bipolar disorder, suicidal intention or attempt
* A score of 6 or more on the 'Ervaringenlijst' (PQ-16) to exclude subclinical susceptibility to psychosis
* Actual abuse of alcohol and/or recreational drugs
* Lifetime history of cardiac valvular disease
* History or evidence of cognitive disorder at screening
* Positive urine drug screen at screening
* Females: Pregnancy, lactation, no acceptable contraceptive use

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-04-16 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in weekly attack frequency, across treatments groups. | week 3 of treatment
  In week 3 post-randomization, compared to the 4-week baseline average per week

SECONDARY OUTCOMES:
Mean change in weekly attack frequency across weeks 4-8 compared to the 4-week baseline and for each week separately. | week 8 post-randomization
100% reduction (remission rate) in number of weekly attacks in the third treatment week, compared to the 4-week baseline, across treatment groups. | week 3 post-randomization
  Rate of subjects with 100% reduction in weekly attack frequency compared to baseline
≥50% reduction (50% responder rate) in number of weekly attacks in the third treatment week, compared to the 4-week baseline, across treatment groups. | week 3 post-randomization
  Rate of subjects with more than 50% reduction in weekly attack frequency compared to baseline
≥30% reduction (30% responder rate) in number of weekly attacks in the third treatment week, compared to the 4-week baseline, across treatment groups. | week 3 post-randomization
  Rate of subjects with more than 30% reduction in weekly attack frequency compared to baseline
100% reduction (remission rate) in number of weekly attacks across weeks 4-8 compared to the 4-week baseline and for each week separately. | week 8 post-randomization
  Rate of subjects with 100% reduction in weekly attack frequency compared to baseline
≥50% reduction (50% responder rate) in number of weekly attacks across weeks 4-8 compared to the 4-week baseline and for each week separately. | week 8 post-randomization
  Rate of subjects with 50% reduction in weekly attack frequency compared to baseline
≥30% reduction (30% responder rate) in number of weekly attacks across weeks 4-8 compared to the 4-week baseline and for each week separately. | week 8 post-randomization
  Rate of subjects with 30% reduction in weekly attack frequency compared to baseline
Mean change in weekly attack frequency in the entire 3 week treatment period compared to the 4-week baseline. | week 3 post-randomization
Mean change in mean headache attack duration (minutes) per week, across treatment groups | week 3 post-randomization
  In week 3 compared to the weekly average during 4-week baseline
Mean change in mean headache attack duration (minutes) per week, across treatment groups | week 8 post-randomization
  Across weeks 4-8 compared to the 4-week baseline and for each week separately.
Mean change in mean headache attack severity (VAS 1-10), across treatment groups | week 3 post-randomization
  In week 3 compared to the weekly average during 4-week baseline
Mean change in mean headache attack severity (VAS 1-10), across treatment groups | week 8 post-randomization
  Across weeks 4-8 compared to the 4-week baseline and for each week separately.
Mean change in number of abortive medication use, across treatment groups | week 3 post-randomization
  In week 3 compared to the weekly average during 4-week baseline
Mean change in number of abortive medication use, across treatment groups | week 8 post-randomization
  Across weeks 4-8 compared to the 4-week baseline
Failure of sustained response' | Weeks 4-8 post-randomization
  Time to initiation of additional prophylactic treatment and/or GON-block during weeks 4-8, across treatment groups
Patient Global Impression of Change (PGIC) | Day 21 post-randomization
  Patient Global Impression of Change at week 3 post-randomization; scale 0-7, higher scores representing better improvement
Patient Global Impression of Change (PGIC) | weeks 3 and 8
  Patient Global Impression of Change at week 8 post-randomization; scale 0-7, higher scores representing better improvement
Health-related quality of life | weeks 3 and 8
  Change from baseline in EQ-5D-5L Visual Analogue Scale (VAS) at weeks 3 and 8.
Hospital Anxiety and Depression Score (HADS) | weeks 3 and 8.
  Change from baseline in Hospital Anxiety and Depression Scale (HADS) at weeks 3 and 8.
Pharmacokinetic (PK)-pharmacodynamic (PD) modelling | Day 18 post-randomization
  Plasma LSD concentrations on day 18 post-randomization frequency
Cost-effectiveness analysis (CEA) from a societal perspective comparing the LSD intervention with usual care. | Week 1, 3 and 8
  Healthcare use and productivity losses will be measured by patient questionnaires (iMCQ, and iPCQ)
Efficacy of treatment masking | Week 1 and 3 post-randomization
  measured as perceived treatment assignment on a 5-point scale (likely verum/possibly verum/don't know/possibly placebo/likely placebo).

OTHER OUTCOMES:
Alcohol consumption | during the entire 12-week duration of the study
  Units of alcohol consumed during baseline, treatment and follow-up
PK-PD modelling | Week 1 and 3
  Correlation between individual pharmacokinetics of LSD and relative change of weekly attack frequency

CONTACTS AND LOCATIONS:
Overall Officials: Kees Kramers, Prof., Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center (LUMC), Leiden
  - Canisius-Wilhelmina Ziekenhuis (CWZ), Nijmegen

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data underlying publication, after deidentification, will be shared upon request to the corresponding author
Supporting Information: Study Protocol
Time Frame: 9-36 months after article publication
Access Criteria: For purpose of meta-analysis and approved by an independent review board

REFERENCES:
- [Background] Hoffmann J, May A. Diagnosis, pathophysiology, and management of cluster headache. Lancet Neurol. 2018 Jan;17(1):75-83. doi: 10.1016/S1474-4422(17)30405-2. Epub 2017 Nov 23. PMID 29174963
- [Background] Rozen TD, Fishman RS. Cluster headache in the United States of America: demographics, clinical characteristics, triggers, suicidality, and personal burden. Headache. 2012 Jan;52(1):99-113. doi: 10.1111/j.1526-4610.2011.02028.x. Epub 2011 Nov 11. PMID 22077141
- [Background] Tepper SJ, Stillman MJ. Cluster headache: potential options for medically refractory patients (when all else fails). Headache. 2013 Jul-Aug;53(7):1183-90. doi: 10.1111/head.12148. Epub 2013 Jun 28. PMID 23808603
- [Background] McGeeney BE. Cannabinoids and hallucinogens for headache. Headache. 2013 Mar;53(3):447-58. doi: 10.1111/head.12025. Epub 2012 Dec 20. PMID 23278122
- [Background] Andersson M, Persson M, Kjellgren A. Psychoactive substances as a last resort-a qualitative study of self-treatment of migraine and cluster headaches. Harm Reduct J. 2017 Sep 5;14(1):60. doi: 10.1186/s12954-017-0186-6. PMID 28870224
- [Background] Sewell RA, Halpern JH, Pope HG Jr. Response of cluster headache to psilocybin and LSD. Neurology. 2006 Jun 27;66(12):1920-2. doi: 10.1212/01.wnl.0000219761.05466.43. PMID 16801660
- [Background] Schindler EA, Gottschalk CH, Weil MJ, Shapiro RE, Wright DA, Sewell RA. Indoleamine Hallucinogens in Cluster Headache: Results of the Clusterbusters Medication Use Survey. J Psychoactive Drugs. 2015 Nov-Dec;47(5):372-81. doi: 10.1080/02791072.2015.1107664. Epub 2015 Nov 23. PMID 26595349
- [Background] de Coo IF, Naber WC, Wilbrink LA, Haan J, Ferrari MD, Fronczek R. Increased use of illicit drugs in a Dutch cluster headache population. Cephalalgia. 2019 Apr;39(5):626-634. doi: 10.1177/0333102418804160. Epub 2018 Oct 5. PMID 30290701